CLINICAL TRIAL: NCT06760130
Title: Retrospective Evaluation of Infections After Delivery
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: INFPP_2022
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-11

CONDITIONS: Postpartum Infection
Keywords: ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In general, transabdominal and transvaginal ultrasound represent the first imaging method in the study of suspected postpartum infections because of its good sensitivity, low cost, and high safety for patients (in fact, it allows the patient to be studied at the bedside, even in clinically unstable patients, it is well tolerated by patients, and it has no risks). CT has an excellent sensitivity in the diagnosis of postpartum infections, however, it has some drawbacks: it is not an examination that can be performed in clinically unstable patients, it cannot be performed at the patient's bedside, it has high costs, and it involves the administration of a significant dose of radiation . There are conflicting data in the literature regarding which examination is most useful for the diagnosis/management of infections in postpartum. Therefore, the investigators want to evaluate whether ultrasound alone, compared with management with combined ultrasound and CT scan, is a useful and sufficient diagnostic tool for the diagnosis and management of postpartum infectious complications.

DETAILED DESCRIPTION:
Cases of infection recorded as a result of these parts will be reviewed. Laboratory tests and clinical data of these will be reviewed. Instrumental, ultrasound and CT images taken in the postpartum for diagnostic confirmation and subsequent follow-up will also be reviewed.

For each patient, information will be collected on:

* Age, weight, height
* Previous pregnancies and their outcome
* Pregnancy that arose spontaneously or through Medically Assisted Procreation techniques
* Conditions concomitant or complicating pregnancy
* Pregnancy outcome (spontaneous delivery or cesarean section)
* Laboratory tests
* Clinical data collected during hospitalization (vital parameters, symptoms, any medications administered)
* Radiologic (CT) or ultrasound (transabdominal and/or transvaginal) investigations performed during the hospital stay, in continuation-iter or in a subsequent hospitalization: name and model (and probe, for ultrasound examinations) of the equipment used will be specified for each examination performed.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older
* Diagnosis of postpartum infection (within 30 days after delivery).

Clinical diagnosis is established by the following criteria (two or more of the following):

* Temperature >38°C or <36°C
* HR >100 bpm
* FR >20 respiratory acts/min or PaCO2 <32mmHg
* GB >14 x 109/dL or <4 x 109/dL
* EGA: lactates >2mmol/L (or 18 mg/dL)
* PCR >2DS from normal value
* Procalcitonin >2DS from normal value or positive laboratory culture result for the presence of bacteria (urinoculture, peritoneal fluid culture, abscess...).
* obtaining informed consent
* Women who have had at least one ultrasound (transabdominal and/or transvaginal) and one CT scan for suspected postpartum infection

Exclusion Criteria:

* Women with localized or systemic infection following infection unrelated to delivery or incision site (in case of cesarean section), such as pneumonia, mastitis, influenza, COVID-19.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: It is planned to enroll patients who gave birth at the Operative Unit of Obstetrics and Prenatal Age Medicine of IRCCS AOUBO Policlinico di Sant'Orsola from 01/01/2017 to 31/12/2021.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of ultrasound signs of infection on ultrasonography | Within 90 days after delivery
  Presence of a hypoanechogenic area at the fascial level or hyperechogenic echoes at the level of the endometrial cavity. Ultrasound signs will be compared with CT scans of patients with established postpartum infection. CT scans are currently the gold standard for the diagnosis of infection, and investigators will rely on what is in the report in the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Brunelli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy